CLINICAL TRIAL: NCT04658017
Title: Feasibility of Hemodialysis With the GARNET Device in Chronic Hemodialysis Patients With a Bloodstream Infection
Brief Title: GARNET™ Filter (GARNET Device) IDE Used in Chronic Hemodialysis Patients With a Bloodstream Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boa Biomedical, Inc. (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 700-00002
Record Dates: First submitted 2020-11-19; First posted 2020-12-08 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Bloodstream Infection
Keywords: Dialysis; Blood Stream Infection; Infection; Bloodstream; PAMPs; Hemodialysis; Sepsis
MeSH Terms: conditions — Sepsis; Infections

STUDY DESIGN:
Intervention Model Description: All enrolled subjects will receive treatment with the GARNET device
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- GARNET device (Experimental): All enrolled subjects will receive treatment with the GARNET device.
  Interventions: Device: GARNET device

INTERVENTIONS:
Device: GARNET device — Use of new filter in conjunction with standard of care dialysis.

SUMMARY:
To evaluate the feasibility of performing combined hemodialysis with the GARNET device in chronic hemodialysis patients with a blood stream infection (BSI), and measure clinical performance and safety endpoints.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single- arm study. Each subject will receive two (2) sessions of hemodialysis with the GARNET each of 3-4 hour duration at a blood flow rate of 250 to 400 mL/min. Any necessary dialysis treatment dosing prescription changes will be made by the treating physician, based on results of small molecule clearance (i.e., urea reduction ratio (URR)). After the second treatment session with the GARNET device, the subjects will resume their hemodialysis regimen using a standard hemodialyzer. Subjects will be followed for 30 days after the final treatment session to evaluate safety.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized adults (age ≥ 18 years and ≤ 90 years)
2. Patients on chronic hemodialysis for ≥ 3 hours per treatment and a minimum of 3 times per week schedule
3. Suspected or confirmed BSI as defined by:

   a. For a suspected central-line (temporary or tunneled central venous catheters) and non- central line (arterio-venous fistula and arterio-venous graft) vascular infection:

   i. presence of at least one of the following signs or symptoms:

1. fever (>38.0°C), 2. pain*, 3. erythema*, or 4. heat at involved vascular site* (*with no other recognized cause); or

ii. presence of purulent drainage/pus at the vascular site, in accordance with the CDC/NHSN Surveillance Definitions for Specific Types of Infections

b. For other suspected infections:

i. presence of at least 2 of the 4 SIRS criteria:

1. Body temperature > 101°F (38.3°C) or < 96.8°F (36°C);
2. Heart rate > 90 beats per minute;
3. Respiratory rate > 20 breaths per minute;
4. White blood cell count > 12,000/mm³, < 4,000/mm³, or > 10% bands

   c. For confirmed infections:

   i. laboratory-confirmed BSI based on the isolation of an organism from blood cultures; or

   ii. If a laboratory-confirmed BSI due to a commensal organism, the presence of at least one of the following signs or symptoms will be required: fever (>38.0˚C), chills, or hypotension.

4. Subject agrees to comply with all follow-up evaluations

5. Subject has provided written informed consent; or if unable to perform informed consent, written informed consent on behalf of the subject has been provided by a legally-authorized representative.

Exclusion Criteria:

1. Pregnancy confirmed by positive urine or serum test, or lactating mothers
2. Subject with severe concomitant disease expected to prolong hospitalization or cause death in ≤ 30 days, or terminal illness, or "do not resuscitate" code status
3. Known sensitivity/allergy to heparin
4. Known sensitivity/allergy to polyethersulfone dialyzers
5. Active bleeding (e.g. active GI bleeding, hematuria or epistaxis, untreated coagulopathy or bleeding from a non-compressible site)
6. Severe thrombocytopenia (platelet count < 50,000/μL)
7. Active enrollment in another study (patients enrolled in an observational study without any interventions or in post-market surveillance do not need to be excluded)
8. Inability to achieve vascular access blood flow rates of ≥250mL/min during the previous dialysis treatment
9. Requirement for Continuous Renal Replacement Therapy/Sustained Low Efficiency Dialysis (CRRT/SLED) due to hemodynamic instability
10. Hemodynamic instability
11. Medical conditions requiring regular blood transfusion
12. Hypocalcemia or clinical symptoms of hypocalcemia at time of enrollment
13. History of or known hypercoagulable state (e.g. Systemic Lupus Erythematosus (SLE), antiphospholipid syndrome/lupus anticoagulant, protein C or S deficiency, antithrombin deficiency, factor V Leiden deficiency, active cancer, sickle cell disease, and history of deep vein thrombosis (DVT))
14. History of a condition documented in the medical record within 6 months prior to enrollment that may result in an increased risk for thrombosis, including any of the following:

    1. Multiple incidents (≥ 2) of unresolvable thrombosis-induced catheter malfunctions which required catheter exchange, occurring within the 6 months prior to enrollment
    2. Prior history of renal transplant thrombosis
    3. Elevated Factor VIII with or without familial hypercholesterolemia
    4. Hyperhomocysteinemia with a homocysteine level of >4 mg/L (17.2 μmol/L)
15. Currently taking oral contraception

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-10-15 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety - Rate of adjudicated device- or GARNET device procedure-related Serious Adverse Events (SAEs) | 30-day follow-up post-2nd GARNET device treatment
  Rate of adjudicated device or GARNET device procedure-related Serious Adverse Events (SAEs) All primary safety endpoints will be reported as adjudicated by the designated Clinical Events Committee (CEC) during treatment and through the 30-day follow-up period.

SECONDARY OUTCOMES:
Resolution of Blood Stream Infection at 30-days post 2nd GARNET device treatment | 30-day follow-up post-2nd GARNET device treatment
  • Resolution of Blood Stream Infection
Clearance for small (blood urea nitrogen) and middle (beta-2-microglobulin) molecule solutes by the GARNET device, as measured by the intra-dialytic urea and beta-2-microglobulin reduction ratio. | During Week 1 participation - Day 0: pre and post first GARNET device treatment and pre and post second GARNET device treatment which must occur by Day 7.
  • Extent of clearance of solutes (small and middle molecules)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - George Washington University, Washington D.C., District of Columbia
  - University of Maryland at Baltimore, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Oregon Health and Science University, Portland, Oregon
  - Houston Methodist, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.